CLINICAL TRIAL: NCT00879918
Title: Pharmacogenetics of Nicotine Metabolism in African-Americans
Acronym: 5075-AAPK1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10-00208; NIDA DA002277
Record Dates: First submitted 2009-04-09; First posted 2009-04-13 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-05

CONDITIONS: Cigarette Smoking
Keywords: Cigarette Smoking in African Americans
MeSH Terms: conditions — Cigarette Smoking | interventions — Cotinine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nicotine pharmacokinetics (Experimental): circadian smoking protocol and IV pharmacokinetic protocol
  Interventions: Drug: Deuterated nicotine and cotinine

INTERVENTIONS:
Drug: Deuterated nicotine and cotinine — used as a marker for pharmacokinetic studies

SUMMARY:
The investigators hypothesize that African Americans (AAs) smoke more for positive reinforcement from nicotine with a "peak-seeking" pattern of smoking (smoking individual cigarettes more intensively with greater intake of nicotine and tobacco smoke toxins), while whites smoke more for negative reinforcement with a "trough-maintaining" pattern (avoiding withdrawal by maintaining more consistent nicotine levels throughout the day by means of a more regular smoking pattern). The investigators believe that these patterns are linked to identifiable racial differences in nicotine pharmacology and that there will be associated racial differences in responses to pharmacologic interventions.

DETAILED DESCRIPTION:
Smoking is the major preventable cause of cancer, premature cardiovascular disease and chronic obstructive lung disease, reproductive problems and infections. AA smokers have a substantially higher risk of cancer and reproductive disorders compared to whites. A recently published large cohort study (183,000 subjects) found a two-fold higher incidence of lung cancer in AAs compared to whites (at cigarette consumption levels of <10 and 11-20 CPD, but not for >30 CPD) (1).

Several lines of evidence indicate that AAs are more highly addicted to cigarette smoking than are whites. AAs are more likely to smoke their first cigarette within 10 minutes of awakening, an indicator of the severity of the dependence.(2) They are more likely to want to quit smoking and are more likely to try to quit (attempts lasting at least 24 hours),(3) but are significantly less likely than whites to be successful abstainers at one year. The quit ratio (former smokers/ever smokers) was recently reported to be 37.3% in AAs compared to 51% for whites.(2)

Research suggests that AAs, who smoke fewer CPD but take in more nicotine per cigarette, are behaving like peak-seekers (smoking primarily for the direct nicotine-mediated positive reinforcement). In contrast, whites, who smoke more CPD with less nicotine intake per cigarette, are behaving more like trough-maintainers (seeking to maintain consistent nicotine levels through the day, presumably to avoid withdrawal symptoms and/or to desensitize receptors).

Studies in our laboratory have shown that AAs metabolize nicotine, and to a greater extent, cotinine, more slowly than do whites (7,10) with slower metabolism by both the CYP2A6 and glucuronidation pathways. We have used the 3HC/COT ratio measured in blood or urine in several studies to show that CYP2A6 activity is lower in AAs compared to whites, including among children. More than 90 CYP2A6 gene variants have been identified. Although many are uncommon and their activity has not been determined (12), some are associated with large individual differences in the rate of nicotine metabolism (13). Studies of CYP2A6 genetics in AAs have only recently been reported. It is unclear whether reported gene variants in AAs can explain the substantial differences in nicotine and especially cotinine metabolism that we have observed in our prior studies. A comprehensive study of nicotine and cotinine kinetics and metabolism after IV dosing in relation to genotype, such as we have recently conducted in whites, is proposed to understand the metabolism of nicotine in AAs.

ELIGIBILITY:
Inclusion Criteria:

* African-American
* Age 18-65
* Smoke at least 5 cigarettes per day

Exclusion Criteria:

* Significant health conditions
* Drug use
* Pregnancy or breastfeeding
* Inability to read English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Nicotine clearance | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Neal L Benowitz, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco/SFGH, San Francisco, California, United States